CLINICAL TRIAL: NCT06523504
Title: Efficacy and Safety of Low-concentration Atropine Eye Drops (0.02%, 0.04%) Combined With Defocus Incorporated Multiple Segments (DIMS) for Moderate and High Myopia Control
Brief Title: Atropine (0.02%, 0.04%) Combined With Defocus DIMS for Moderate and High Myopia Control
Acronym: atropine
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ruihua Wei (Other)
Collaborators: Beijing Tongren Hospital (Other)
Responsible Party: Sponsor-Investigator, Ruihua Wei, Professor, Tianjin Medical University Eye Hospital
Organization: Tianjin Medical University Eye Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019yj001J-5; 2019yj001J-5 (Other Grant/Funding Number: Beijing Bethune Charitable Foundation)
Record Dates: First submitted 2024-07-19; First posted 2024-07-26 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- The DIMS Group (Experimental): wear DIMS ,and use placebo,once nightly, both eye
  Interventions: Device: DIMS
- 0.02% ATP (Experimental): wear SP, and use 0.02%ATP eye drops, once nightly, both eye
  Interventions: Drug: The 0.02% ATP Group
- 0.04%ATP (Experimental): wear SP, and use 0.04%ATP eye drops, once nightly, both eye
  Interventions: Drug: The 0.04% ATP Group
- 0.02%ATP+DIMS (Experimental): wear DIMS, and use 0.02%ATP eye drops, once nightly, both eye
  Interventions: Combination Product: 0.02%ATP+DIMS
- 0.04%ATP+DIMS (Experimental): wear DIMS, and use 0.04%ATP eye drops, once nightly, both eye
  Interventions: Combination Product: 0.04%ATP+DIMS

INTERVENTIONS:
Device: DIMS — wear DIMS ,and use placebo,once nightly, both eye
  Arms: The DIMS Group
Drug: The 0.02% ATP Group — wear SP, and use 0.02%ATP eye drops, once nightly, both eye
  Arms: 0.02% ATP
Drug: The 0.04% ATP Group — wear SP, and use 0.04%ATP eye drops, once nightly, both eye
  Arms: 0.04%ATP
Combination Product: 0.02%ATP+DIMS — wear DIMS, and use 0.02%ATP eye drops, once nightly, both eye
  Arms: 0.02%ATP+DIMS
Combination Product: 0.04%ATP+DIMS — wear DIMS, and use 0.04%ATP eye drops, once nightly, both eye
  Arms: 0.04%ATP+DIMS

SUMMARY:
To evaluate the effectiveness and safety of DIMS, low concentration atropine eye drops,and atropine combined with DIMS in controlling axial length and refraction in children with moderate to high myopia.

DETAILED DESCRIPTION:
In this study, stratified block randomization was employed for random grouping, and the total sample size required as calculated was 410 individuals. Firstly, 410 subjects were assigned ID numbers ranging from 1 to 410. SPSS.26 statistical software was utilized to apply the "random number generator" by setting the "fixed seed number" to "20231121", and subsequently generate random numbers. Once the random numbers were obtained, random sampling and grouping were conducted. This study was a multicenter trial, with block randomization stratified by center. The total sample size of 410 was distributed across 4 cities, and the samples collected in each city were randomly allocated into 5 treatment groups (groups A, B, C, D, and E), with approximately 20 individuals in each group.

ELIGIBILITY:
Inclusion Criteria:

* School-age children aged 6 to 12 years (including boundary value)
* Children with moderate or high myopia (subjective refraction after cycloplegia: -9.00D≤spherical equivalent (SE)≤-3.00D, with-rule astigmatism (C)≤2.00D, against-rule astigmatism (C)≤1.00D, anisometropia of both eyes≤2.50D)
* Binocular best corrected visual acuity (BCVA)≥0.8 (five-point visual acuity 4.9)
* Agree with the study scheme and sign the informed consent
* Note: if both eyes meet the inclusion criteria, the eye with higher spherical equivalent is the study eye; if one eye meets the inclusion criteria, the eye is the study eye.

Exclusion Criteria:

* Used or currently using orthokeratology, multifocal contact lenses, defocusing framework lenses, atropine eye drops and other myopia control means in the past month; used red light treatment in the past
* Children with obvious strabismus and amblyopia
* With congenital eye disease, such as congenital cataract, congenital retinal disease
* Secondary myopia (such as premature retinopathy or other eye diseases in infants and children caused secondary myopia), or myopia combined with systemic syndrome (such as Marfan syndrome)
* Had internal eye surgery (such as cataract extraction, intraocular lens implantation, anti-glaucoma surgery, etc.)
* Refractive medium opacity (such as corneal disease, crystal opacity, etc.)
* Bnormal intraocular pressure and clinical significance (IOP <10 mmHg or IOP >21mmHg or binocular IOP difference ≥5mmHg)
* Fundus chorioretinopathy (except for high myopia fundus degenerative changes) or other intraocular diseases
* Optic nerve damage or congenital optic nerve dysfunction
* Can not be regularly checked
* The adjustment range is less than 8D or obvious near difficulties
* Other reasons researchers think it is not suitable for inclusion in researchers

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 410 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Best Corrected Visual Acuity | up to 24 months
  Best Corrected Visual Acuity

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Eye Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No